CLINICAL TRIAL: NCT03100461
Title: Adaptive Intervention to Maximize Colorectal Screening in Safety Net Populations
Acronym: AIMSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00002929; 1R01CA188898-01A1 (NIH)
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2020-05

CONDITIONS: Colorectal Cancer
Keywords: Cancer Screening; Colon Cancer; Colon Cancer Screening
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HE + HE (Active Comparator): Participants receive up to two interventions. Participants receive HE initially and then a second time if not screened after 6 months.
  Interventions: Other: Health Education
- HE + I2 (Active Comparator): Participants receive up to two interventions. Participants receive HE initially and then I2 if not screened after 6 months.
  Interventions: Other: I2; Other: Health Education
- I2 + I2 (Experimental): Participants receive up to two interventions. Participants receive I2 initially and then a second time if not screened after 6 months.
  Interventions: Other: I2
- I2 + HE (Active Comparator): Participants receive up to two interventions. Participants receive I2 initially and then HE if not screened after 6 months.
  Interventions: Other: I2; Other: Health Education

INTERVENTIONS:
Other: I2 — A touch screen computer delivered "implementation intentions" (I2) intervention on CRC screening. "Implementation intentions" are the exact steps (the when, what, where, how) one will take to complete a test (the date and time, at home or at the doctor's office, with what supplies, etc.).
  Other Names: Implementation Intentions
  Arms: HE + I2; I2 + HE; I2 + I2
Other: Health Education — Standard of care approach that will provide basic information on CRC screening.
  Arms: HE + HE; HE + I2; I2 + HE

SUMMARY:
The goal of this study is to find the best ways to increase colorectal cancer (CRC) screening.

DETAILED DESCRIPTION:
Colorectal Cancer is preventable and curable but is still the second most common cause of cancer death in the U.S. Minorities and those with low income have more CRC than middle and high income Whites.. They also get fewer CRC screening tests. Low knowledge of CRC screening may, in part, drive this lower test use. We need new ways to improve CRC screening in primary care clinics where many minority and uninsured patients receive health care.

ELIGIBILITY:
Inclusion Criteria:

* Have a home address and access to a working telephone
* Pass Mini-Cog assessment

Exclusion Criteria:

* FIT (fecal immunochemical test) test within 1 year, Sigmoidoscopy or Barium enema within 5 years, or Colonoscopy within 10 years
* Acute medical illness,
* current GI bleed
* history of adenomatous polyps
* Colorectal Cancer
* 1st degree relative with CRC < age 60 years
* inherited polyposis/non-polyposis syndrome
* inflammatory bowel disease
* Another household member enrolled in the study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
CRC screening completion rate | 12-14 Months
  Rate of participants who receive CRC screening during study participation

SECONDARY OUTCOMES:
Cost analysis of each intervention pathway | 14 Months
  Measure will be calculated by estimating all cost factors in the CRC screening process, include personnel and materials/supplies costs, materials development costs, and time of all study staff involved. Measure represented as a per participant cost to complete screening.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Greiner, MD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States